CLINICAL TRIAL: NCT05712798
Title: Physiological Responses to Exercise Tests in Primary Ciliary Dyskinesia Compared With Healthy Children and Investigation of the Relationship Between Exercise Capacity and Quality of Life in Primary Ciliary Dyskinesia
Brief Title: Physiological Responses to Exercise Tests in Primary Ciliary Dyskinesia Compared With Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Principal Investigator, Hacettepe University
Other Study IDs: GO 20/647
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The children with primary ciliary dyskinesia: The children with primary ciliary dyskinesia
  Interventions: Other: No intervention
- Healthy controls: Healthy children
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The individuals with primary ciliary dyskinesia (PCD) have lower aerobic fitness and anaerobic performance than healthy individuals. Cardiopulmonary exercise test (CPET) provides an integrated assessment of integrative exercise responses involving the pulmonary, cardiovascular, hematopoietic, neuropsychological, and skeletal muscle systems that are not adequately reflected by measurement of the function of organ systems. Maximum oxygen consumption is measured by performing gas exchange analysis with CPET, offering an objective measure of cardiorespiratory fitness. The six-minute walk test (6MWT) and the shuttle walk test (SWT) are field tests that produce oxygen consumption results similar to those during CPET. There is a need to determine the physiological responses to CPET, SWT and 6MWT in individuals with PCD. Additionally, the physiological responses of individuals with PCD to different exercise tests will be compared with the responses of healthy individuals. Low aerobic capacity in individuals with PCD may affect the physical, emotional, and social lives of individuals. This influence may cause a decrease in the quality of life of individuals with PCD. The relationship between exercise capacity and quality of life in individuals with PSD will be investigated with this study.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with PCD in the Pediatrics Department, Pediatric Chest Diseases Unit of Hacettepe University Faculty of Medicine and being routinely referred to Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit for physiotherapy applications and pulmonary rehabilitation program,
* Being clinically stable,
* Being between 8-18 years old,
* Having a forced expiratory volume in the first second (FEV1) ≥ 40%,

The healthy group will be composed of individuals who do not have any known disease and volunteer to participate in the study. For healthy individuals, volunteers from acquaintances and/or relatives of the researchers will be included in the study.

Exclusion Criteria:

* Having unstable clinical condition
* Having severe neuromuscular and musculoskeletal problems,
* Having any congenital heart diseases other than situs inversus,
* Unable to cooperate

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The children with primary ciliary dyskinesia and healthy children
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
Shuttle walk test distance | up to 3 weeks
  Shuttle walk test distance will be determined using shuttle walk test
Quality of life score | 1st day
  Quality of life score will be determined using multidimensional measure to assess health-related quality of life in primary ciliary dyskinesia (QoL-PCD).
Maximal oxygen uptake | up to 3 weeks
  Maximal oxygen uptake will be determined using cardiopulmonary exercise test.
6 minute walk test distance | up to 3 weeks
  6 minute walk test distance will be determined using 6 minute walk test

SECONDARY OUTCOMES:
Pulmonary function test - forced vital capacity | 1st day
  Pulmonary function test using a spirometer will be performed. Forced vital capacity will be recorded.
Pulmonary function test - Forced expiratory volume in one second | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second will be recorded.
Maximal inspiratory pressure | 1st day
  Maximal inspiratory pressure will be measured using a mouthpiece device.
Maximal expiratory pressure | 1st day
  Maximal expiratory pressure will be measured using a mouthpiece device.
Pulmonary function test - Peak expiratory flow | 1st day
  Pulmonary function test using a spirometer will be performed. Peak expiratory flow will be recorded.
Pulmonary function test - Forced mid-expiratory flow (FEF25-75) | 1stday
  Pulmonary function test using a spirometer will be performed. Peak expiratory flow will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, Study Chair — Hacettepe University; Ugur Ozcelik, Principal Investigator — Hacettepe University; Nagehan Emiralioglu, Principal Investigator — Hacettepe University; Melda Saglam, Principal Investigator — Hacettepe University; Naciye Vardar-Yagli, Principal Investigator — Hacettepe University; Ebru Calik-Kutukcu, Principal Investigator — Hacettepe University; Birce Sunman, Principal Investigator — Hacettepe University; Hazal Sonbahar-Ulu, Principal Investigator — Akdeniz University; Aslihan Cakmak, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cakmak-Onal A, Kocaaga E, Sonbahar-Ulu H, Calik E, Vardar-Yagli N, Saglam M, Sunman B, Emiralioglu N, Ozcelik U, Inal-Ince D. Physiological responses to cardiopulmonary and field exercise tests in primary ciliary dyskinesia compared with healthy peers. Eur J Appl Physiol. 2025 Nov 4. doi: 10.1007/s00421-025-06019-2. Online ahead of print. PMID 41186743